CLINICAL TRIAL: NCT05409508
Title: Psychological Management by Meditation of Full COnscience in Virtual REality of People With Amyotrophic Lateral Sclerosis: Effects on Cognition, Behavior, Quality of Life and Psychological Well-being
Acronym: COREVALS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-A01230-43
Record Dates: First submitted 2022-05-30; First posted 2022-06-08 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-05

CONDITIONS: Lateral Sclerosis Amyotrophy; Mindfulness Meditation
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with mindfulness meditation care (Experimental)
  Interventions: Other: mindfulness meditation care
- Patients without mindfulness meditation care (Active Comparator)
  Interventions: Other: no mindfulness meditation care

INTERVENTIONS:
Other: mindfulness meditation care — mindfulness meditation care
  Arms: Patients with mindfulness meditation care
Other: no mindfulness meditation care — no mindfulness meditation care
  Arms: Patients without mindfulness meditation care

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a neurodegenerative disease that results in progressive paralysis of the muscles involved in voluntary motor skills, speech, swallowing and breathing. It also causes non-motor symptoms including psychological, cognitive and behavioral difficulties that have a negative impact on patients' quality of life, well-being and long-term development. There is no curative therapy for ALS and drug treatments have little effect on non-motor symptoms. Interventions based on mindfulness meditation, defined as a state of consciousness that arises when one decides to focus attention in the present moment without judgment on the real experience, seem to be a promising tool for the reduction of non-motor symptoms in a number of progressive neurological conditions (Alzheimer's disease, multiple sclerosis, etc.), suggesting that mindfulness significantly helps in the management of these symptoms. Our project therefore aims to implement a mindfulness meditation program adapted to the management of non-motor symptoms in ALS based on virtual reality (VR).

ELIGIBILITY:
Inclusion Criteria:

* Majors to inclusion
* Mother tongue: French
* Patients for whom ALS of bulbar or spinal form defined according to El Escorial criteria is possible, probable or certain
* Able to carry out the investigations and interventions provided for in the protocol
* Signature of informed consent to participate in the study

Exclusion Criteria:

* Participation in intervention research modifying management
* History likely to disrupt cognition (constituted stroke, sequelae of traumatic brain injury, active epilepsy, learning disabilities, alcohol dependence syndrome, drug use, psychiatric disorders), severe cognitive impairment (MMSE <24)
* People who meet the diagnostic criteria for Frontotemporal Dementia
* Pregnant or lactating women
* Persons deprived of their liberty by administrative or judicial decision
* Persons undergoing psychiatric care under duress
* Persons subject to a legal protection measure
* Persons unable to express their consent
* Persons not affiliated or not beneficiaries of a social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
To assess the benefits of psychological care with mindfulness meditation in virtual reality versus psychological management without mindfulness meditation in virtual reality in terms of evolution over time | at 3 months
  from a quality of life scale : ALSSQOL-R : the lower the score, the more the person feels a sense of well-being